CLINICAL TRIAL: NCT03787667
Title: Application of Radiomics in Precise Preoperative Diagnosis and Prognsis Evaluation of Colorectal Cancer: a Prospective, Clinical Study
Brief Title: Application of Radiomics in Precise Preoperative Diagnosis and Prognsis Evaluation of Colorectal Cancer.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Guoxiang Cai, Professor, Fudan University
Other Study IDs: ColoRadiomics
Record Dates: First submitted 2018-12-22; First posted 2018-12-26 (Actual); Last update posted 2018-12-26 (Actual); Status verified 2018-12

CONDITIONS: Colorectal Cancer Stage I-IV
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with pathologically diagnosed colorectal cancer: Patients with pathologically diagnosed colorectal cancer
  Interventions: Diagnostic Test: CT or MRI based Radiomics

INTERVENTIONS:
Diagnostic Test: CT or MRI based Radiomics — Radiomic features were extracted from enhanced CT or MRI of colorectal cancer.

SUMMARY:
This is a prospective, clinical study. This study is to collect and analyze data of radiomics of primary site or metastasis of colorectal cancer aiming to precisizing preoperative diagnosis and long-term prognsis evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pathologically confirmed colorectal cancer
* Male or female aged 18-75 years old on the day of signing informed consent.
* Patients who received imageological examination of primary or metastasis
* Patients who received surgical resection of primary or metastasis
* Patients must have a performance status of ≤1 on the ECOG Performance Scale.
* Colorectal cancer is the only malignant tumor
* Written informed consent must be obtained from patient or patient's legal representative and ability for patient to comply with the requirements of the study

Exclusion Criteria:

* Patients received adjuvant treatment prior to imageological examination
* Tis stage patients
* Paitents who diagnosed with malignant disease within 5 years.
* Patients with a history or current evidence of any condition or abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study, or is not in the best interest of the patient to participate, in the opinion of the Investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients received enhaced CT or MRI test must have baseline evaluations performed prior to the study and must meet all inclusion and exclusion criteria. In addition, the patient must be thoroughly informed about all aspects of the study, including the study visit schedule and required evaluations and all regulatory requirements for informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity | 2 years
  The sensitivity of radiomics in predicting regional or distant synchronous colorectal metastasis

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China